CLINICAL TRIAL: NCT02365779
Title: Dynamic Real-time in Vivo Confocal Laser Endomicroscopy Cellvizio® of the Fallopian Tube During Laparoscopy
Brief Title: Optical Biopsy and Fallopian Tube
Acronym: FALLOPTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014.875
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Bilateral Laparoscopic Salpingectomy
Keywords: salpingectomy; optical biopsy; Cellvizio®

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bilateral laparoscopic salpingectomy (Experimental)
  Interventions: Procedure: bilateral laparoscopic salpingectomy; Device: endomicroscopy Cellvizio® system

INTERVENTIONS:
Procedure: bilateral laparoscopic salpingectomy — Use of the confocal laser endomicroscopy Cellvizio® system during laparoscopy salpingectomy
Device: endomicroscopy Cellvizio® system

SUMMARY:
High-grade serous ovarian cancer is the most threatening type of gynaecological cancer with an important mortality due to late diagnosis. However the prognosis is excellent in the early stages of the disease. Recently it has been described a new serous carcinogenic sequence from the fallopian tube with tubal precancerous lesions. Therefore the identification of these early preinvasive lesions would be of great interest in the population with hereditary predisposition for ovarian cancer (concept of oncofertility) and in the general population (to determine whether bilateral salpingectomy has to be performed during a hysterectomy for benign disease).

The optical biopsy has been developed and validated in the detection of early precancerous lesions (such as Barrett's oesophagus or in situ cancer of the bladder). The first objective of this study is to prospectively assess the efficacy of optical biopsy (Cellvizio®) in the study of fallopian tubes during laparoscopy with correlation between the histopathological and immunohistochemical analysis and the endomicroscopy image interpretation. The second objective is to describe the optical biopsy pictures in order to state a classification.

DETAILED DESCRIPTION:
Inclusion Criteria:

* Woman aged 18 years or more
* All patients with laparoscopic salpingectomy for benign conditions (tubal ligation, during a hysterectomy), for prophylactic conditions (BRCA mutation) or in case of pelvic cancers
* Informed and signed consent

Exclusion Criteria:

* Interview revealing disorder entailing unacceptable risk of postoperative complications: coagulation disorder, immune system disorder, evolutive disease, etc.
* Pregnancy, ongoing or planned during the study period
* Allergy to fluorescein
* Previous allergy or anaphylactic shock during an angiography
* Allergic or hypersensibility reactions
* Severe asthma, chronic cardiac or pulmonary diseases
* Restricted renal function
* Patient under a beta-blockers treatment
* Inability to understand information provided
* Not covered by a national health insurance scheme, prisoner or under administrative supervision

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18 years or more
* All patients with laparoscopic salpingectomy for benign conditions (tubal ligation, during a hysterectomy), for prophylactic conditions (BRCA mutation) or in case of pelvic cancers
* Informed and signed consent

Exclusion Criteria:

* Interview revealing disorder entailing unacceptable risk of postoperative complications: coagulation disorder, immune system disorder, evolutive disease, etc.
* Pregnancy, ongoing or planned during the study period
* Allergy to fluorescein
* Previous allergy or anaphylactic shock during an angiography
* Allergic or hypersensibility reactions
* Severe asthma, chronic cardiac or pulmonary diseases
* Restricted renal function
* Patient under a beta-blockers treatment
* Inability to understand information provided
* Not covered by a national health insurance scheme, prisoner or under administrative supervision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Correlation between the histopathological and immunohistochemical analysis and the endomicroscopy image interpretation | DAY 1

SECONDARY OUTCOMES:
: Description of the optical biopsy pictures in order to state a classification | DAY 1

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie, Hôpital Femme Mère Enfant, Lyon, Bron, France

REFERENCES:
- [Background] Chene G, Chauvy L, Buenerd A, Moret S, Nadaud B, Beaufils E, Le Bail-Carval K, Chabert P, Mellier G, Lamblin G. In vivo confocal laser endomicroscopy during laparoscopy for gynecological surgery: A promising tool. J Gynecol Obstet Hum Reprod. 2017 Sep;46(7):565-569. doi: 10.1016/j.jogoh.2017.06.003. Epub 2017 Jun 23. PMID 28652089
- [Background] Chene G, Chauvy L, Buenerd A, Moret S, Nadaud B, Chabert P, Lamblin G. Dynamic real-time in vivo confocal laser endomicroscopy of the fallopian tube during laparoscopy in the prevention of ovarian cancer. Eur J Obstet Gynecol Reprod Biol. 2017 Sep;216:18-23. doi: 10.1016/j.ejogrb.2017.07.002. Epub 2017 Jul 5. PMID 28692889